CLINICAL TRIAL: NCT02322996
Title: Phenotyping Acute Pain for Discovery Research and Directed Therapeutics
Status: Withdrawn | Type: Observational
Why Stopped: never started
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Raymond Dionne, Raymond A. Dionne, DDS, PhD Research Professor Department of Pharmacology & Toxicology Brody School of Medicine Department of Foundational Sciences School of Dental Medicine East Carolina University Greenville, NC 27834-4354, East Carolina University
Other Study IDs: 14-001670
Record Dates: First submitted 2014-12-10; First posted 2014-12-23 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Post op Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- open label: After the surgery and the onset of moderate-severe pain, QST and PROMIS questionnaires will be repeated. Throughout these procedures, patients will rate their pain perception using a numeric rating scale. Approximately 2-3 hours after surgery at the onset of moderate pain, the rescue analgesic (toradol) will be administered via intramuscular injection. Again, QST and PROMIS protocols will be repeated after the drug is given and when patients report pain relief. A standard naproxen dose of 500 mg will be given to patients upon leaving the clinic and they will be instructed to take one pill orally each day before returning for evaluation after 48 hours.
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — The deep phenotyping of acute pain will be conducted using the oral surgery model. Before surgery, subjects will undergo QST and answer short-form questionnaires related to pain and activities of daily living.

SUMMARY:
The goal of the current study is to combine existing and new tools for quantifying patient self-report to characterize changes in acute pain. The ability to quantitatively measure self-report provides behavioral pain phenotypes that can serve as the basis for clustering patients into sub-groups based on their self-report of their symptoms, eliminating observer based perceptions of patients' pain.

DETAILED DESCRIPTION:
Pain is a therapeutic challenge as well as a public health problem that is estimated to affect over 116 million American adults [1]; reduces quality of life; and is estimated to cost up to $635 billion annually. Growing recognition of the need for evidence-based, individual-centered treatment strategies raises expectations that health care will be improved by matching proven effective treatments with knowledge of patients' unique characteristics to optimize efficacy and safety. Essential to the goal of matching treatments to patients to enhance analgesic drug development and therapy is identification of intermediate phenotypes that capture the mechanistic complexity, genetic expression and epigenetic changes of hundreds of ongoing processes and mediators that influence treatment efficacy and safety and may form the basis for differential responses to drug therapy. The ability to identify functional variants in the genomic responses to pain and therapeutics at the sub-group and patient levels, however, has been limited to date by lack of thorough phenotyping for patients with pain.

The need for a more comprehensive understanding of human phenotypes has spawned a new method of phenotyping studies referred to as "deep phenotyping." Deep phenotyping for pharmacogenomic studies requires both breath and depth to better interpret the complexities of genomic variations that may underlie individual differences in pain report. One approach to address this complexity is to use quantitative testing of clinical features to identify more homogeneous subsets within a group of patients with a given diagnosis or characteristic. Variations in quantitative measures may identify intermediate phenotypes that are genetically less complex yet have potentially stronger signals closer to the site of gene action. In pain, quantitative testing is often termed "quantitative sensory testing", or QST.

Exclusion

1. Current or history of mental disorder or substance abuse
2. Allergy to aspirin, NSAIDS, or sulfonamide
3. Pregnant and/or nursing
4. History of peptic ulcers and/or GI bleeding
5. Concurrent use of agents which may obscure pain report, e.g., alcohol, opioids, benzodiazepines, and depressants, etc
6. Chronic use of medications confounding assessment of the inflammatory response or analgesia, e.g., antihistamines, NSAIDS, steroids, antidepressants
7. Concurrent or history of chronic diseases, e.g., diabetes, rheumatoid arthritis, liver disease, cancer, hypertension or obesity (body mass index >35)
8. Expectation of excessive surgical difficulty, resulting in a difficulty score of 5 for any tooth (determined from panoramic radiograph)
9. Subjects with extreme anxiety and who are candidates for general anesthesia or conscious sedation

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 and older willing to undergo clinically indicated non-emergent oral surgery for the removal of impacted third molars with local anesthesia
2. Indicated for the removal of third molars, at least a minimum of one partial-bony impacted third molar, with a total difficulty score total of not less than 4*
3. Communicate in spoken and written English
4. Willing to undergo research observation for 4 hours postoperatively and 48 hour follow up visit
5. In good health with an ASA status of 1 or 2 by self report and review of medical history
6. Self-report of moderate or severe pain on a categorical scale with a minimum of 4 out of 10 on the numerical rating scale following the offset of local anesthesia

   * 1=erupted, 2=soft tissue impaction, 3=partial bony impaction, 4=full bony impaction, 5 = unusual surgical difficulty

Exclusion Criteria:

1. Current or history of mental disorder or substance abuse
2. Allergy to aspirin, NSAIDS, or sulfonamide
3. Pregnant and/or nursing
4. History of peptic ulcers and/or GI bleeding
5. Concurrent use of agents which may obscure pain report, e.g., alcohol, opioids, benzodiazepines, and depressants, etc
6. Chronic use of medications confounding assessment of the inflammatory response or analgesia, e.g., antihistamines, NSAIDS, steroids, antidepressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male or females over 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
characterize changes in acute pain | 48 hours
  The goal of the current study is to combine existing and new tools for quantifying patient self-report to characterize changes in acute pain

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Dionne, DDS, Principal Investigator — School of Dental Medicine at East Carolina University
Locations (1):
- School of Dental Medicine At East Carolina University, Greenville, North Carolina, United States